CLINICAL TRIAL: NCT01195168
Title: Assessment of Cardiovascular Risk in PCOS-a Cross Sectional Study of Women With PCOS Compared With Controls Matched for Age, Body Mass Index and, or Insulin Resistance
Brief Title: Cardiovascular Risk Markers in Polycystic Ovary Syndrome (PCOS)
Acronym: CS
Status: Completed | Type: Observational
Sponsor: The Adelaide and Meath Hospital (Other)
Collaborators: University College Dublin (Other)
Responsible Party: Dr James Gibney, The Adelaide and Meath Hospital Incorporating the National Children's Hospital
Other Study IDs: DDC-UCD-CS
Record Dates: First submitted 2010-09-02; First posted 2010-09-06 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2008-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PCOS cohort: Women with PCOS as diagnosed by the NIH criteria
- Control cohort: Women without PCOS

SUMMARY:
Women with polycystic ovary syndrome (PCOS) are more often overweight or obese and are more insulin resistant than women without the condition and may be at greater risk of developing cardiovascular disease. It is not know whether it is the overweight and insulin resistant component of PCOS, or PCOS per se which leads to the greater cardiovascular disease risk. The aim of this study was to examine cardiovascular risk markers in women with PCOS versus a control population matched for body mass index (BMI), and or, insulin resistance

ELIGIBILITY:
Inclusion Criteria:

* Had a positive diagnosis of PCOS as defined according to the NIH criteria as chronic oligomenorrhoea (< 9 menstrual cycles per year) and clinical and/or biochemical evidence of hyperandrogenism, in the absence of other disorders causing the same phenotype. Clinical criteria included hirsutism with a Ferriman-Galwey score greater than 9, acne or male pattern alopecia; biochemical criteria included total-testosterone, androstenedione or dehydroepiandrosterone sulphate (DHEAS) greater than the laboratory reference range.
* Were between the ages of 18 and 40

Exclusion Criteria:

* Were under 18 years or greater than 40 years old,
* Were non-Caucasian
* Were pregnant, lactating or trying to conceive
* Had a body mass index (BMI) <18kg/m2 or >50kg/m2
* Had a recent illness or any chronic illness likely to influence results
* Were taking hormonal contraception

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with PCOS and a control population of women matched for age and body mass index (BMI) and insulin resistance
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2006-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Assessment of Insulin resistance in women with PCOS compared with BMI and age matched controls | Recruitment ran from Nov 2006-July 2008; Each subject attended the study location fasting on one occasion
  Subjects underwent a standard 75g oral glucose tolerance test (OGTT) and blood were taken fasting and at 2 hours. Surrogate markers of insulin resistance (HOMA) and insulin sensitivity (Avignon index of Insulin Sensitivity; QUICKI) were calculated

SECONDARY OUTCOMES:
Assessment of concentrations of androgens in women with PCOS compared with controls | Recruitment ran from Nov 2006-July 2008; Each subject attended the study location fasting on one occasion
  Bloods were taken in the fasted state and circulating concentrations of androgens (DHEAS, testosterone, androstenedione) were assessed
Assessment of lipid profile in women with PCOS compared with age matched controls | Recruitment ran from Nov 2006-July 2008; Each subject attended the study location fasting on one occasion
  Bloods were taken in the fasted state and circulating concentrations of lipids assessed
Assessment of inflammatory profile in women with PCOS compared with controls | Recruitment ran from Nov 2006-July 2008; Each subject attended the study location fasting on one occasion
  Bloods were taken in the fasted state and circulating concetrations of several important markers of inflammation as well as key adipokines were assessed

CONTACTS AND LOCATIONS:
Overall Officials: James Gibney, Dr, Principal Investigator — The Adelaide and Meath Hospital; Helen M Roche, Prof, Principal Investigator — University College Dublin
Locations (2):
- Ireland (2):
  - Diabetes Day Centre, The Adelaide and Meath Hosptial, Dublin, Leinster
  - Nutrigenomics Research Group, University College Dublin, Dublin, Leinster

REFERENCES:
- [Derived] Gidwani S, Phelan N, McGill J, McGowan A, O'Connor A, Young IS, Gibney J, McEneny J. Polycystic ovary syndrome influences the level of serum amyloid A and activity of phospholipid transfer protein in HDL(2) and HDL(3). Hum Reprod. 2014 Jul;29(7):1518-25. doi: 10.1093/humrep/deu115. Epub 2014 May 19. PMID 24842896
- [Derived] Phelan N, O'Connor A, Kyaw Tun T, Correia N, Boran G, Roche HM, Gibney J. Hormonal and metabolic effects of polyunsaturated fatty acids in young women with polycystic ovary syndrome: results from a cross-sectional analysis and a randomized, placebo-controlled, crossover trial. Am J Clin Nutr. 2011 Mar;93(3):652-62. doi: 10.3945/ajcn.110.005538. Epub 2011 Jan 26. PMID 21270384